CLINICAL TRIAL: NCT02311803
Title: Preservation Versus Excision of Denonvilliers Fascia in Laparoscopic Pelvic Autonomic Nerve Preserving Surgery for Male Mid-low Rectal Cancer Patients: a Randomized Controlled Clinical Trial
Brief Title: Preservation Versus Excision of Denonvilliers Fascia in L-PANP Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongbo Wei, Assistant to the Dean, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PED-PANP001
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

ARMS (2):
- Preservation of Denonvilliers Fascia (Experimental): Preservation of Denonvilliers Fascia in Laparoscopy-assisted pelvic autonomic nerve preservation surgery for male mid-low rectal cancer patients
  Interventions: Procedure: Preservation of Denonvilliers Fascia
- Excision of Denonvilliers Fascia (Active Comparator): Excision of Denonvilliers Fascia in Laparoscopy-assisted pelvic autonomic nerve preservation surgery for male mid-low rectal cancer patients
  Interventions: Procedure: Excision of Denonvilliers Fascia

INTERVENTIONS:
Procedure: Preservation of Denonvilliers Fascia — In this group, patients accepte L-PANP surgery without excision of Denonvilliers Fascia
  Arms: Preservation of Denonvilliers Fascia
Procedure: Excision of Denonvilliers Fascia — In this group, patients accepte L-PANP surgery with excision of Denonvilliers Fascia
  Arms: Excision of Denonvilliers Fascia

SUMMARY:
TME (Total mesorectum excision) is the golden standard of radical resection for mid-low rectal cancer. However, the damage of pelvic autonomic nerve following with TME principle will lead to high incidence of urinary and sexual function disorder. PANP (pelvic autonomic nerve preservation) surgery played a role in decreasing incidence of urinary and sexual function disorder. However, 32%-44% patients still suffered from urinary and sexual function disorder when underwent open (O-PANP-TME) or laparoscopic PANP TME surgery (L-PANP-TME).

In the early stage of work, the investigators performed preservation of Denovilliers' fascia in L-PANP-TME to discuss the protection of urinary and sexual function of male mid-low rectal cancer patients. The results showed that preservation of Denovilliers' fascia in L-PANP-TME significantly decreased incidence of urinary and sexual function disorder. In order to further confirm the early work, the investigators design a randomized controlled clinical trial to compare differences in urinary and sexual function protection and long-term outcomes between preservation and excision of Denovilliers' fascia in L-PANP-TME.

ELIGIBILITY:
Inclusion Criteria:

1. Age from over 20 to under 60 years;
2. Primary rectal adenocarcinoma confirmed pathologically by endoscopic biopsy;
3. Mid-low rectal cancer (distance from anal edge≤12cm);
4. cT1-3, N0-3, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual Seventh Edition;
5. Expected curative resection through L-PANP;
6. Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale;
7. ASA (American Society of Anesthesiology) score class I, II, or III;
8. Written informed consent;
9. Urinary and sexual function normal preoperatively

Exclusion Criteria:

1. Severe mental disorder;
2. History of previous pelvic surgery;
3. Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging;
4. History of other malignant disease within past five years;
5. History of unstable angina or myocardial infarction within past six months;
6. History of cerebrovascular accident within past six months;
7. History of continuous systematic administration of corticosteroids within one month;
8. Contraindication of heart, brain, lung, etc dysfunction;
9. Requirement of simultaneous surgery for other disease;
10. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by rectal cancer;
11. Rectal cancer invades surrounding tissues;
12. Existence of genuine incontinence or severe stress incontinence preoperatively

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 172 (Estimated)
Dates: Start 2015-02; Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Urinary function | 30 days
  Urodynamic study and IPSS (International prostate symptom score) are used to assess urinary function
Sexual function | 30 days
  IIEF-5 (International questionnaire of erectile function-5) and Ejaculation function classification are used to assess sexual function
3-year disease free survival rate | 36 months
5-year disease free survival rate | 60 months
Urinary function | 36 months
  Urodynamic study and IPSS (International prostate symptom score) are used to assess urinary function
Sexual function | 36 months
  IIEF-5 (International questionnaire of erectile function-5) and Ejaculation function classification are used to assess sexual function

SECONDARY OUTCOMES:
Morbidity | 30 days
3-year overall survival rate | 36 months
3-year recurrence pattern | 36 months
Mortality | 30 days
Morbidity | 36 months
Mortality | 36 months
5-year overall survival rate | 60 months
5-year recurrence pattern | 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China